CLINICAL TRIAL: NCT02841241
Title: Esmolol to Control Adrenergic Storm in Septic Shock - Roll-in
Brief Title: Esmolol Infusion for Patients With Septic Shock and Persistent Tachycardia
Acronym: ECASSS-R
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1050147
Record Dates: First submitted 2016-07-14; First posted 2016-07-22 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Septic Shock
Keywords: esmolol; adrenergic storm; septic shock
MeSH Terms: conditions — Shock, Septic | interventions — esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Esmolol (Experimental): Esmolol infusion, started without bolus, with slow upward titration to a maximum infusion rate is protocolized, with a target heart rate of 80-90/min
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Esmolol — Esmolol infusion
  Other Names: Brevibloc

SUMMARY:
This is a prospective, single arm, "roll-in" study of esmolol infusion for patients with septic shock with persistent tachycardia after adequate intravenous volume expansion. The study will evaluate the adequacy and efficiency of study protocols for the anticipated, main ECASSS study, which will have a separate entry in clinicaltrials.gov.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To evaluate the adequacy and efficiency of study protocols for the anticipated, randomized, controlled ECASSS study. The primary clinical outcome is organ-failure free days at 28 days, with multiple secondary outcomes, including those relevant to function of and compliance with the study protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Within 48 hours of admission to the ICU and septic shock (sepsis present at time of admission)

   a. Septic shock defined by consensus criteria as i. At least two systemic inflammatory response syndrome (SIRS) criteria ii. Suspected or documented infection iii. Receiving vasopressors to treat hypotension after at least 20 ml/kg intravenous crystalloid volume expansion
3. Receiving vasopressors through a central venous catheter for more than 60 minutes.
4. Arterial catheter in place or expected to be placed imminently.
5. Heart rate > 90/min while receiving vasopressors for more than 60 minutes.
6. Adequately volume expanded, as manifest by any of the following, performed as part of routine clinical care (i.e., no study procedures will be performed before signed consent). If none of these measures are clinically available, the clinical attending must confirm that volume expansion is adequate. (After enrollment, a final safety check will confirm the adequacy of volume expansion.)

   1. Central venous pressure (CVP) > 15 mm Hg.
   2. Negative Passive-Leg Raise (PLR) maneuver (<10% increase in cardiac output after PLR).
   3. No cardiac output response (<10% increase) after rapid infusion (<5 min) of 250 ml of IV crystalloid, i.e., a graded volume expansion challenge (GVEC).
   4. For patients who happen to be breathing passively on a positive pressure mechanical ventilator delivering at least 8 ml/kg tidal volumes and in normal sinus rhythm, stroke volume variability <10% (such patients are acknowledged to be uncommon; the protocol does not recommend or require the induction of passive breathing).

Exclusion Criteria:

1. Lack of informed consent.
2. Currently receiving ECMO (extracorporeal membrane oxygenation).
3. Known pregnancy or nursing.
4. Patient is a prisoner.
5. Patient on hospice (or equivalent comfort care approach) at or before the time of enrollment.
6. Known or current atrial fibrillation.
7. Previously enrolled in the trial.
8. Known allergy to esmolol or vehicle
9. Receipt of nodal blocking agents within three half lives
10. Hemoglobin < 7 gm/dl.
11. Cardiac arrest within 24 hours.
12. Pulmonary hypertension (moderate or severe), from documented history of prior right heart catheterization or current evidence on TTE (transthoracic echocardiography) of any of the following

    * mPAP (mean pulmonary artery pressure) ≥ 35 mmHg
    * SPAP (systolic pulmonary artery pressure)≥ 60 mmHg
13. Cardiovascular collapse, as manifested by inability to achieve a MAP (mean arterial pressure) of 65 mmHg with vasopressor therapy.
14. Cardiogenic shock, as defined by any of the following

    * Cardiac index ≤ 2 L/min/m2
    * Ejection fraction ≤ 25%
    * ScvO2 ≤ 60%
    * Current infusion of any dose of dobutamine, milrinone, or dopamine
    * Current infusion of epinephrine for clinically diagnosed cardiogenic shock
15. Significant atrioventricular dysfunction

    * Sick sinus syndrome
    * PR interval (time from onset of P wave to start of QRS complex) > 200 msec
    * Current evidence or prior history of Grade 2 or Grade 3 heart block
    * Pacemaker or plans to place a pacemaker
16. Pheochromocytoma or status asthmaticus
17. Receiving clonidine, guanfacine, or moxonidine
18. Hemoglobin < 7 gm/dl
19. Cardiovascular collapse (failure to achieve MAP of 65mmHg)
20. Cardiac arrest within 24 hours
21. Worse than moderate aortic stenosis

    • Known aortic stenosis, with any of (1) mean gradient ≥ 40 mmHg OR (2) maximum gradient ≥ 60mmHg OR (3) aortic valve area ≤ 1.0cm2 OR (4) aortic valve area index ≤ 0.85cm2/m2 body surface area.
22. Worse than mild mitral stenosis • Known mitral stenosis, with any of (1) valve area ≤ 1.5 cm2 OR mean gradient ≥ 5 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Brown, MD,MS, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center and Intermountain Clinics, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudiger A, Singer M. The heart in sepsis: from basic mechanisms to clinical management. Curr Vasc Pharmacol. 2013 Mar 1;11(2):187-95. PMID 23506497
- [Background] Novotny NM, Lahm T, Markel TA, Crisostomo PR, Wang M, Wang Y, Ray R, Tan J, Al-Azzawi D, Meldrum DR. beta-Blockers in sepsis: reexamining the evidence. Shock. 2009 Feb;31(2):113-9. doi: 10.1097/SHK.0b013e318180ffb6. PMID 18636043
- [Background] Oberbeck R, Kobbe P. Beta-adrenergic antagonists: indications and potential immunomodulatory side effects in the critically ill. Curr Med Chem. 2009;16(9):1082-90. doi: 10.2174/092986709787581770. PMID 19275613
- [Background] Morelli A, Ertmer C, Westphal M, Rehberg S, Kampmeier T, Ligges S, Orecchioni A, D'Egidio A, D'Ippoliti F, Raffone C, Venditti M, Guarracino F, Girardis M, Tritapepe L, Pietropaoli P, Mebazaa A, Singer M. Effect of heart rate control with esmolol on hemodynamic and clinical outcomes in patients with septic shock: a randomized clinical trial. JAMA. 2013 Oct 23;310(16):1683-91. doi: 10.1001/jama.2013.278477. PMID 24108526
- [Derived] Brown SM, Beesley SJ, Lanspa MJ, Grissom CK, Wilson EL, Parikh SM, Sarge T, Talmor D, Banner-Goodspeed V, Novack V, Thompson BT, Shahul S; Esmolol to Control Adrenergic Storm in Septic Shock-ROLL-IN (ECASSS-R) study. Esmolol infusion in patients with septic shock and tachycardia: a prospective, single-arm, feasibility study. Pilot Feasibility Stud. 2018 Aug 3;4:132. doi: 10.1186/s40814-018-0321-5. eCollection 2018. PMID 30123523
- See also: Esmolol infusion in patients with septic shock and tachycardia: a prospective, single-arm, feasibility study — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-018-0321-5

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Esmolol
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Esmolol
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Admission APACHE (Acute Physiologic Assessment and Chronic Health Evaluation) II [Mean (Standard Deviation); unit: Units on a scale (0-100)] — "estimates ICU mortality based on a number of laboratory values and patient signs taking both acute and chronic disease into account"; score is from 0-100, with 0 being a low risk of mortality and 35-100 being a high risk
  Units on a scale (0-100) | 28 (8)

OUTCOME MEASURES:

1. Primary Outcome: Organ-failure-free Days
Description: As of day 28, the number of calendar days on which the patient receives none of (a) vasopressor therapy, (b) mechanical ventilation, or (c) renal replacement therapy. If the patients dies on or before day 28, they have -1 organ-failure-free days.
  The resulting point-based score combines the probability of death and the number of days without organ failure.
  Score of -1 = Death before day 28 (Lowest Score). Score of 28 = Patient has been successful at going 28 without any vasopressor therapy/mechanical ventilation/renal replacement therapy (Highest Score)
Time Frame: Day 28
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Esmolol
Number analyzed (Participants) | 7
units on a scale | 26 [24.5 to 26]

2. Secondary Outcome: All-cause Mortality
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Esmolol
Number analyzed (Participants) | 7
Participants | 0

3. Secondary Outcome: Peak Serum High-sensitivity Troponin
Description: Measured after enrollment.
Time Frame: Troponin is measured on day 0 and day 1 (first day of esmolol infusion is day 0)
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Esmolol
Number analyzed (Participants) | 7
ng/ml | 0.14 [0.12 to 0.47]

4. Secondary Outcome: Left Ventricular Global Longitudinal Strain at 24 Hours
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: Percentage of myocardial shortening (%)
Arm/Group | Esmolol
Number analyzed (Participants) | 7
Percentage of myocardial shortening (%) | -15.8 [-20.1 to -13.5]

5. Secondary Outcome: Development of Heart Block
Time Frame: for duration of esmolol infusion, an expected average of 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Esmolol
Number analyzed (Participants) | 7
Participants | 0

6. Other Pre Specified Outcome: Proportion of Compliance With Final Safety Check
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Esmolol
Number analyzed (Participants) | 7
Participants | 7

7. Other Pre Specified Outcome: Percentage Hourly Checks During Which Protocol Compliance Was Observed
Description: For the esmolol titration protocol, each hour (the closest value of heart rate to the hour) during the esmolol infusion will be determined to be "in range" or "out of range," with 3bpm margin for compliance (i.e., heart rate 77 to 93bpm). The initiation and cessation of esmolol will also be included as a timepoint for evaluation of compliance. Protocol compliance is considered adequate where overall compliance on hourly checks is >80%.
Time Frame: for duration of esmolol infusion, an expected average of 2 days
Measure: Mean (Standard Deviation); unit: Percentage of hourly checks
Arm/Group | Esmolol
Number analyzed (Participants) | 7
Percentage of hourly checks | 98 (4.4)

8. Other Pre Specified Outcome: Number of Participants With Intolerance to Esmolol Infusion at Any Given Rate
Description: Patients who met a prespecified stop event for esmolol titration, suggesting intolerance to a given infusion rate.
  Per protocol, study drug titration: "The target heart rate is 85 bpm. Start study drug infusion at 20 mcg/kg/min, without bolus, if HR (heart rate) ≥ 100 bpm. If HR >90 bpm and <100 bpm, start study drug infusion at 10 mcg/kg/min, without bolus. Increase by 20 mcg/kg/min every 20 minutes as long as HR > 90 bpm, to a maximum dose of 100 mcg/kg/min. If HR < 80 bpm and > 70 bpm, decrease infusion rate by 10 mcg/kg/min; if HR ≤ 70 bpm and > 60 bpm, decrease infusion rate by 20 mcg/kg/min."
Time Frame: duration of esmolol infusion (~2 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Esmolol
Number analyzed (Participants) | 7
Participants | 3

ADVERSE EVENTS:
Time Frame: Duration of esmolol infusion (approximately 2 days)
Arm/Group | Esmolol
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT02841241/Prot_SAP_ICF_000.pdf